CLINICAL TRIAL: NCT02563080
Title: Development of Pancreatic Exocrine Insufficiency After Moderately Severe or Severe Acute Pancreatitis
Brief Title: Pancreatic Exocrine Insufficiency in Acute Pancreatitis
Acronym: APPEI
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Leena Kylanpaa, MD, PhD, Helsinki University Central Hospital
Other Study IDs: Exocrine insufficiency
Record Dates: First submitted 2015-09-27; First posted 2015-09-29 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Exocrine Pancreatic Insufficiency; Acute Pancreatitis
Keywords: exocrine insufficiency; acute pancreatitis; severe; moderately severe
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: None Retained — Fecal samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First attack of acute pancreatitis: 50 patients with first attack of moderately severe or severe acute pancreatitis treated in Helsinki University Hospital.

SUMMARY:
Severe pancreatitis induces more damage in the pancreas and might therefore result reduced exocrine function leading to the insufficiency. The aim of this prospective study is to investigate development of pancreatic exocrine insufficiency in patients recovering from first attack of moderately severe or severe acute pancreatitis.

DETAILED DESCRIPTION:
This is a prospective pilot study of 50 patients with first attack of moderately severe or severe acute pancreatitis (AP) classified by the new revised criteria for AP 2012 treated in Helsinki University Hospital. The included patients are treated according to the existing hospital practice and current guidelines for AP (American Pancreatic Association guidelines). The development of pancreatic exocrine insufficiency is determined by measuring the fecal elastase-1 test. The test is measured during the hospitalization time (baseline testing), and in the follow-up period 1-2 months and 12 months after discharging from hospital. The baseline test will be measured as soon as the severity of AP is known and patient is included in the study, and the first stool sample is available. Patients with previous history of AP, chronic pancreatitis, known pancreatic exocrine insufficiency or previous pancreatic surgery will be excluded.

The patients' characteristics (age, gender, comorbidities) and etiology of AP, laboratory values on admission, imaging findings and data of given treatments and interventional therapies and length of hospital stays are collected from hospital charts. Also the 30-day and hospital mortality will be recorded. Patients' symptoms (weight loss, diarrhea, abdominal pain) and BMIs are recorded with physical examinations in the 1-2 months follow-up visit. 12 months after discharging from hospital the patients' symptoms and BMIs are recorded with phone inquiries. 5-year survival after the first AP attack will be determined from hospital records.

The approval of the ethics committee of the hospital has been obtained. An informed consent will be obtained from all patients.

Development of pancreatic exocrine insufficiency after first attack of moderately severe or severe AP confirmed by fecal elastase-1 test is the primary endpoint of this study. Also, the persistence pancreatic exocrine insufficiency and probable new developments of it during the follow-up will be assessed (secondary endpoints). 30-day and hospital mortality and 5-year survival after first attack of moderately severe or severe AP will be determined as well (secondary endpoints).

The aim in this study (during the study period) is not to change the existing management of AP. The existing guidelines for treatment of severe AP patients do not include enzyme supplementation therapy. However, if the patients have low fecal elastase-1 levels indicating pancreatic exocrine insufficiency after the follow-up period of 12 months, they will be informed about the enzyme supplementation therapy. And if the patients are willing to start the therapy, it can be administrated.

ELIGIBILITY:
Inclusion Criteria:

* first episode of acute pancreatitis (diagnosis based on acute onset of characteristic symptoms and elevated plasma levels of amylase and/or typical findings on CT)
* severity of acute pancreatitis classified as moderately severe or severe by revised Atlanta classification of acute pancreatitis 2012

Exclusion Criteria:

* previous history of acute pancreatitis
* chronic pancreatitis
* known pancreatic exocrine insufficiency
* previous pancreatic surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with first attack of moderately severe or severe acute pancreatitis treated in Helsinki University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Development of pancreatic exocrine insufficiency after first attack of moderately severe or severe acute pancreatitis confirmed by fecal elastase-1 test. | One year after discharging from hospital
  fecal elastase-1 <200 ug/g

SECONDARY OUTCOMES:
Persistence of pancreatic exocrine insufficiency after first attack of moderately severe or severe acute pancreatitis | One year after discharging from hospital
  fecal elastase-1 <200 ug/g
New developments of pancreatic exocrine insufficiency after first attack of moderately severe or severe acute pancreatitis during the follow-up time | One year after discharging from hospital
  fecal elastase-1 <200 ug/g

OTHER OUTCOMES:
30-day and hospital mortality after first attack of acute pancreatitis | 30 days, hospitalization time
  mortality
5-year survival after first attack of acute pancreatitis | 5 years
  survival

CONTACTS AND LOCATIONS:
Overall Officials: Leena Kylänpää, MD,PhD, Principal Investigator — Helsinki University Central Hospital; Outi Lindström, Md,PhD, Study Chair — Helsinki University Central Hospital; Taija Korpela, MD, Study Chair — Helsinki University Central Hospital; Marianne Udd, MD,PhD, Study Chair — Helsinki University Central Hospital; Panu Mentula, MD,PhD, Study Chair — Helsinki University Central Hospital; Päivi Siironen, MD,PhD, Study Chair — Helsinki University Central Hospital; Matti Tolonen, MD, Study Chair — Helsinki University Central Hospital; Elina Lietzen, MD, Study Chair — Turku University Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Boreham B, Ammori BJ. A prospective evaluation of pancreatic exocrine function in patients with acute pancreatitis: correlation with extent of necrosis and pancreatic endocrine insufficiency. Pancreatology. 2003;3(4):303-8. doi: 10.1159/000071768. PMID 12890992
- [Derived] Lindstrom O, Lietzen E, Mentula P, Tolonen M, Siironen P, Udd M, Puolakkainen P, Kylanpaa L. Development of pancreatic exocrine insufficiency after first moderately severe or severe acute pancreatitis. Scand J Gastroenterol. 2025 Sep;60(9):921-927. doi: 10.1080/00365521.2025.2533337. Epub 2025 Jul 17. PMID 40673865